CLINICAL TRIAL: NCT06588608
Title: A Pilot Study of Auricular Vagus Nerve Stimulation on Cardiovascular Biomarkers and Glycemic Homeostasis in Persons With Chronic Spinal Cord Injuries
Brief Title: Auricular Vagus Nerve Stimulation (aVNS) in Chronic Spinal Cord Injuries (SCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Daniel Ganzer, Assistant Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20240490
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- aVNS followed by no aVNS in subjects with SCI (Experimental): Auricular vagal nerve stimulation (aVNS) will be provided by a device that is placed around the ear. A low-voltage electrical signal will be given for 30 minutes. In the following visit, subjects will complete all study assessments without the aVNS. Participation will be up to 2 weeks.
  Interventions: Device: auricular nerve stimulation (aVNS); Device: sham aVNS
- no aVNS followed by aVNS in subjects with SCI (Experimental): Subjects will complete all study assessments without the aVNS. In the following visit, Auricular vagal nerve stimulation (aVNS) will be provided by a device that is placed around the ear. A low-voltage electrical signal will be given for 30 minutes. Participation will be up to 2 weeks.
  Interventions: Device: auricular nerve stimulation (aVNS); Device: sham aVNS

INTERVENTIONS:
Device: auricular nerve stimulation (aVNS) — The Spark Sparrow system stimulates the auricular branch of the Vagus nerve using a low-voltage electrical signal comprising a 1 Hz - 150 Hz biphasic square wave with a pulse width of 50s - 750s. Stimulation current is controlled with a maximum voltage of 95 V and 1-5 milliamperes (mA) output current. The device is positioned at the auricular branch of the Vagus nerve on the ear with the outer electrode in front of the ear and the inner electrode into the hollow area of the ear, just above the ear canal. Stimulation will occur for 30 minutes. Participation will last up to 2 weeks and requires 2 separate in-person visits. Each visit will be up to 3 hours.
Device: sham aVNS — The Spark Sparrow system device will be positioned at the auricular branch of the Vagus nerve on the ear with the outer electrode in front of the ear and the inner electrode into the hollow area of the ear, just above the ear canal. Subjects will wear the device for 30 minutes during which no stimulation will be emitted. Participation will last up to 2 weeks and requires 2 separate in-person visits. Each visit will be up to 3 hours.

SUMMARY:
The purpose of this research is to test if Auricular Vagal Nerve Stimulation (aVNS) is safe in persons with spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Chronic (equal or greater to 1 year) motor-complete and incomplete SCI Abbreviated Injury Scale (AIS) of A or B at the C5-T10 levels

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Prisoner
3. Failure to satisfy inclusion criteria
4. Previous bariatric surgery
5. Active implantable devices (such as pacemakers)
6. Skin irritation or damage at the site (ear)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-related Adverse Events (AEs) | Up to 2 weeks
  Safety will be reported as the number of treatment-related AEs assessed by study PI or physician
Number of subjects that complete the study | Up to 2 weeks
  Safety will be determined by number of subjects that complete the two study, visits (in total, two weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D Ganzer, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No